CLINICAL TRIAL: NCT04434534
Title: Effect of Açaí Juçara Consumption on Endothelial Function and Arterial Stiffness in Overwheight or Obese Individuals: A Randomized Clinical Trial
Brief Title: Effect of Açaí Juçara Consumption on Endothelial Function and Arterial Stiffness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5483/18
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Overweight and Obesity
Keywords: Endhothelial function; Anthocyanins; Arterial stiffness; Açaí Juçara
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hipocaloric Diet with Açaí Juçara (Experimental): Individualized diet plans calculated for each participant, reducing 500-1000 daily calories, including 200g of Açaí Juçara (2 pulps).
  Interventions: Dietary Supplement: Hipocaloric Diet with Açaí Juçara
- Hipocaloric Diet (Active Comparator): Individualized diet plans calculated for each participant, reducing 500-1000 daily calories.
  Interventions: Other: Hipocaloric Diet

INTERVENTIONS:
Dietary Supplement: Hipocaloric Diet with Açaí Juçara — Daily consumption of Açaí Juçara pulp (200g) and nutritional adequacy of meals in individualized diet plans calculated for each participant.
  Arms: Hipocaloric Diet with Açaí Juçara
Other: Hipocaloric Diet — Nutritional adequacy of meals in individualized diet plans calculated for each participant.
  Arms: Hipocaloric Diet

SUMMARY:
This study evaluates the consumption of Açaí Juçara pulp in endothelial function and arterial stiffness in overwheight and obese individuals. Half of participants will receive a hipocaloric diet and two Açaí Juçara pulps for daily consumption, while the other half will receive just a hipocaloric diet.

DETAILED DESCRIPTION:
Obesity is the most prevalent nutritional disease and a growing public health problem worldwide. This clinical condition is an established risk factor for cardiovascular diseases.

Açaí Juçara is a brazilian fruit, rich in antioxidants, like anthocyanin. This compound have antioxidative and vasodilatory properties. Prospective studies have shown that the antioxidant present in berries can improve vascular health, like endothelial function, measured by Flow Mediated Dilatation (FMD) and arterial stiffness, measured by Pulse Wave Velocity (PWV).

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle
* Overwheight or obesity "1" diagnostic (BMI >25kg/m² and <35kg/m²)

Exclusion Criteria:

* Alcoolism
* Smoking
* Diagnostic of Diabetes Mellitus or Coronary Artery Disease
* Use of Statin Therapy
* Cardiovascular diseases
* Infectious Disease

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12-10 (Estimated); Study Completion 2020-12-28 (Estimated)

PRIMARY OUTCOMES:
Flow-mediated Dilation (FMD) | 12 weeks
  The non-invasive evaluation of endothelial function in the brachial artery will be performed at the Laboratory of Clinical Investigation of the Institute of Cardiology of Rio Grande do Sul. The images will be captured by a trained professional in the method using ultrasonography equipament with a linear transducer. The acquisition of the image will be through the program Ulead Video Studio (EasyCap). The protocol consist in 1 minute of baseline recording of the arterial flow diameter, followed by 5 minutes of reactive hyperemia (cuff occlusion in the forearm) and then 3 minutes recording after cuff deflation. The exams will be record in a video, and later analyzed through the Cardiovascular Suite software.
  The FMD will be evaluated before the beginning of the diet and after 12 weeks of diet.

SECONDARY OUTCOMES:
Pulse Wave Velocity | 12 weeks
  The calibrated and validated Mobil-O-Graph® portable monitor will be used. This module is connected to a computer to record the brachial pulse wave. It performs pulse wave analysis based on the oscillometric method. The arterial pulsation generates pressure oscillations, which are transmitted to the blood pressure cuff and measured by the transducer to be interpreted by a specific software, recording the pulse wave of the brachial artery and deriving a pulse wave from the aortic arch.
  All measurements will be performed by the same evaluator on the right side of the volunteer. Participants will be instructed to be in 12 hours os fasting.
  The pulse wave velocity will be evaluated before the beginning of the diet and after 12 weeks of diet.

CONTACTS AND LOCATIONS:
Overall Officials: Tainah Ortiz, Principal Investigator — Instituto de Cardiologia
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul/Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No